CLINICAL TRIAL: NCT00996879
Title: Study to Evaluate the Effect of BMS-791325 on the Pharmacokinetics of the CYP3A4 Probe Midazolam Administered Orally in Healthy Subjects
Brief Title: Study to Assess the Effect of BMS-791325 on the Pharmacokinetics of Midazolam in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AI443-006
Record Dates: First submitted 2009-10-14; First posted 2009-10-16 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Hepatitis C
Keywords: Human Volunteers
MeSH Terms: conditions — Hepatitis C | interventions — Midazolam; 8-cyclohexyl-N-((dimethylamino)sulfonyl)-1,1a,2,12b-tetrahydro-11-methoxy-1a-((3-methyl-3,8-diazabicyclo(3.2.1)oct-8-yl)carbonyl)cycloprop(d)indolo(2,1-a)(2)benzazepine-5-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Midazolam + BMS-791325 (Experimental)
  Interventions: Drug: Midazolam; Drug: BMS-791325

INTERVENTIONS:
Drug: Midazolam — Syrup, Oral, 5 mg, Single dose, 2 days
Drug: BMS-791325 — Capsules, Oral, 300 mg, Every 12 hours, 8 days

SUMMARY:
The purpose of this study is to assess the effect of BMS-791325 on the pharmacokinetics of the CYP3A4 Probe Midazolam.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged 18 to 49 years, with BMI of 18-32 kg/m²
* Women who are not of childbearing potential

Exclusion Criteria:

* Women of childbearing potential
* Women who are pregnant, breastfeeding, or unwilling or unable to use an acceptable method of birth control.
* Gastrointestinal disease that may impact the absorption of study drug
* History of any chronic respiratory disease (asthma, COPD)

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameters area under curve (AUC) (TAU), maximum concentration (Cmax) | Within 24 hours of dosing

SECONDARY OUTCOMES:
Safety assessments will be based on medical review of adverse event reports and the results of vital sign measurements, ECGs, physical examination and clinical laboratory tests | On Days 1, 2, 4, 6, 8, 9, and 10

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Wcct Global, Llc, Cypress, California, United States

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx